CLINICAL TRIAL: NCT06605313
Title: First-in-man Feasibility Study of SQ-Kyrin-T Transcatheter Tricuspid Valve Clip Delivery System and Steerable Guide Catheter in Patients With Severe Tricuspid Regurgitation
Brief Title: SQ-Kyrin-T First-in-man Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVRP01-001
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SQ-Kyrin-T Transcatheter Tricuspid Valve Repair System (Experimental): Subjects who received treatment with the experimental device will be included in this arm.
  Interventions: Device: SQ-Kyrin-T Transcatheter Tricuspid Valve Repair System

INTERVENTIONS:
Device: SQ-Kyrin-T Transcatheter Tricuspid Valve Repair System — Transcathether Edge-to-Edge repair for tricuspid regurgitation with SQ-Kyrin-T Transcatheter Tricuspid Valve Repair System.

SUMMARY:
The goal of this clinical trial is to evaluate the performance, operability and reliability of the SQ-Kyrin-T Transcatheter Edge-to Edge Valve Repair System in treating severe tricuspid regurgitation in Chinese population with high or prohibitive risk for conventional surgery; and to provide safety and efficacy data on which subsequent confirmatory trial can be based.

DETAILED DESCRIPTION:
A prospective, multicenter, single-arm feasibility trial to evaluate the performance, operability and reliability of the SQ-Kyrin-T Transcatheter Edge-to Edge Valve Repair System in treating severe tricuspid regurgitation in Chinese population with high or prohibitive risk for conventional surgery.

It plans to enroll 12 qualified patients. The primary endpoint of the study is the postoperative technical success rate. Patients will be seen for follow-up visits at discharge, 30 days, 6 months, and annually through 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Severe or greater (≥3+) tricuspid regurgitation determined by transthoracic echocardiogram despite adequate treatment per applicable standards.
2. NYHA classification of II, III, or IVa.
3. Age ≥ 18 years old, gender not limited.
4. Patient is determined to be at high or prohibitive risk for tricuspid valve surgery, or is determined to be not suitable for open heart surgery by local multidisciplinary cardiac team (with at least one cardiac surgeon and one cardiologist).
5. Patients who understand the purpose of the trial, voluntarily participate and sign an informed consent form, and are willing to undergo relevant examinations and clinical follow-up.
6. Tricuspid valve coaptation defect<2cm.
7. No significant calcification of tricuspid valve leaflets.
8. Tricuspid valve leaflet anatomy suitable for clip implantation, positioning on the leaflets and sufficient reduction in TR.

Exclusion Criteria:

1. Previous tricuspid valve surgery; previous heart transplant; implanted cardiac electronic device.
2. Any cardiovascular interventional procedure within the past 30 days.
3. Patients with other valvular diseases requiring surgical or interventional treatment.
4. Patients with severe large-vessel disease requiring surgical treatment.
5. Echocardiogram indicating the presence of intracardiac masses, thrombus, or vegetations.
6. Severe uncontrolled hypertension (systolic blood pressure [SBP] ≥ 180 mmHg and/or diastolic blood pressure [DBP] ≥ 110 mmHg).
7. Pulmonary artery systolic pressure > 70 mmHg.
8. Moderate to severe or severe mitral regurgitation (≥3+).
9. Active infective endocarditis, active rheumatic heart disease, or rheumatic tricuspid valve disease.
10. Myocardial infarction or known unstable angina within the past 30 days.
11. Severe untreated coronary artery disease.
12. Hemodynamic instability, defined as SBP < 90 mmHg with or without cardiogenic shock, or the need for an intra-aortic balloon pump or other hemodynamic support device.
13. Cerebrovascular accident within the past 3 months.
14. Renal failure requiring dialysis.
15. Patients with a confirmed coagulation disorder or severe coagulation system disease.
16. Patients with clear contraindications to anticoagulant use.
17. History of acute peptic ulcer or gastrointestinal bleeding within the past 3 months.
18. Known allergy to contrast agents or nickel-titanium alloy products.
19. Tricuspid valve stenosis (defined as a tricuspid valve area ≤ 1.0 cm² and/or a mean trans-tricuspid gradient ≥ 5 mmHg).
20. Left ventricular ejection fraction (LVEF) ≤ 20%.
21. Severe chronic obstructive pulmonary disease requiring continuous oxygen therapy.
22. Life expectancy of less than 12 months.
23. Pregnant or breastfeeding women, or women planning to conceive.
24. Patients deemed to have poor compliance or unable to complete the study as required; or other situations in which the investigator considers the subject unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2027-11-24 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | immediately after intervention
  Defined by the following four conditions:
  1. No procedural mortality. 2. Successful delivery, implant, retrieval of the delivery system. 3. Successful devices release. 4. No need for any emergency surgery related to the device or surgical approach.

SECONDARY OUTCOMES:
Incidence of all-cause mortality | 30 days
Incidence of major adverse events | 30 days
  The major adverse event refers to the composite endpoint of death, stroke, myocardial infarction, and cardiovascular surgery due to device- or interventional-related adverse events that occurred since successful transfemoral vein puncture and establishment of atrial septal pathway.
Device success rate | 30 days
  Defined by the following two conditions:
  1. Technical success maintained at day 30. 2. Echocardiographic tricuspid regurgitation reduction at least 1 grade.
Clinical success rate | 30 days
  Defined by following two conditions:
  1. Device success. 2. No major adverse events occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, MD, Ph.D, Principal Investigator — Fuwai Cardiovascular Hospital of Yunnan Province
Locations (1):
- Fuwai Cardiovascular Hospital of Yunnan Province, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No